CLINICAL TRIAL: NCT05751109
Title: Comparison of Infiltration Between the Popliteal Artery and the Capsule of the Knee (IPACK) Block and Adductor Canal Block Combination Versus Epidural Analgesia for Total Knee Arthroplasty
Brief Title: Comparison of IPACK and Adductor Canal Block Combination Versus Epidural Analgesia for Total Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Rasim Onur Karaoglu, Principal Investigator, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Other Study IDs: 681423
Record Dates: First submitted 2022-09-22; First posted 2023-03-02 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Knee Injuries
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ipack+adductor canal block: The 40 patients received ACB + IPACK (Group 1, n = 40),. All patients were evaluated with VAS score for pain recorded at 1h, 8 h, postoperative day (POD) 1 and 3. month after the surgery. The secondary outcome measures assessed were movement time and discharge time.
  Interventions: Procedure: ipack+adduktor kanal
- epidural analgesia: The 40 patients received combine spinal epidural (Group 2, n = 40),. All patients were evaluated with VAS score for pain recorded at 1h, 8 h, postoperative day (POD) 1 and 3. month after the surgery. The secondary outcome measures assessed were movement time and discharge time.
  Interventions: Procedure: ipack+adduktor kanal

INTERVENTIONS:
Procedure: ipack+adduktor kanal — nerve block
  Other Names: kombine epidural

SUMMARY:
To compare the efficacy and complications of IPACK and adductor canal block combination and epidural block in patients who will be operated for knee arthroscopy under spinal anesthesia.

DETAILED DESCRIPTION:
Between 15.08.2022 and 15.04.2023, the patients who will be operated on for knee surgery under spinal anesthesia, older than 18 years of age were included in the study. Demographic characteristics of the patients, comorbidities, ASA scores, mobilization time, amount of postoperative analgesic use, and postoperative pain scores of the 1. 8. 24. hours will be observed. The vas score at the 3rd month was learned over the phone.

ELIGIBILITY:
Inclusion Criteria:

* Those who consented to participate in the study
* Patients over the age of 18 who will be operated on due to knee pathology
* Patients to be operated under spinal anesthesia
* Disease that will limit cooperation

Exclusion Criteria:

* Patients under the age of 18
* Patients to be operated under general anesthesia
* Disease that will cause limited cooperation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 80 people
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-08-16 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) evaluation for postoperative pain | 8. Hour
  The Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) evaluation for postoperative pain | 1. Hour
  The Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').
Visual Analogue Scale (VAS) evaluation for postoperative pain | 24. Hour
  The Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Onur Karaoglu, Istanbul, Kağıthane
  - Rasim Onur Karaoglu, Istanbul, Kağıthane